CLINICAL TRIAL: NCT01176071
Title: An Observational Assessment of the Correlation Between Circulating Galactomannan and Beta-D-glucan and Clinical Outcome in the Setting of Invasive Aspergillosis in Patients With an Underlying Hematological Disorder
Brief Title: Correlation Between Circulating Galactomannan and Beta-D-glucan and Clinical Outcome of Invasive Aspergillosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Maertens Johan, UZ Gasthuisberg Leuven
Other Study IDs: IISP 37367
Record Dates: First submitted 2010-08-04; First posted 2010-08-05 (Estimated); Last update posted 2010-08-05 (Estimated); Status verified 2010-07

CONDITIONS: Invasive Aspergillosis
Keywords: galactomannan; beta-D-glucan; aspergillosis; outcome
MeSH Terms: conditions — Aspergillosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators hypothesize that early galactomannan and beta-D-glucan features, namely the height of the initial value at the time of diagnosis and the subsequent rate of marker decay within the first week(s) following therapy (day 7, day 14) are important factors in predicting clinical outcome.

DETAILED DESCRIPTION:
A major challenge in the development of antifungal therapies for invasive fungal infections is the difficulty in assessing early treatment response and clinical prognosis. Mycological endpoints are often unreliable, reflected by the low sensitivity of fungal cultures to diagnose infection (20% for aspergillosis). Radiographic endpoints can be misleading, particularly when assessed early following treatment initiation. Clinical endpoints can be ambiguous indicators of treatment response, and generally include categorization of patient outcome as better, stable or worse. Furthermore, clinical assessments are likely confounded by the underlying diseases predisposing to fungal infection. Thus, a biomarker interposed between the initiation of antifungal therapy and patient outcome would bring much needed precision in the evaluation of novel antifungal drugs and thus serve as a valuable tool to guide decision-taking regarding ineffective treatments and dose selection in product development. The current absence of such biomarkers represents a critical capability gap. To date, only few studies have examined the prognostic value of fungal biomarkers in invasive aspergillosis on clinical outcome and have been limited by sample seize. To address this issue, the current study will examine the correlation between the fungal biomarkers galactomannan and beta-D-glucan with clinical outcome in invasive aspergillosis. The study will also incorporate C-reactive protein (CRP) levels, as they seem to be a useful surrogate marker of IL-6 production.

The investigator contains a sample database of 100+ patients with either probable or proven invasive aspergillosis for which daily marker levels and CRP (during the first two weeks of antifungal therapy) were measured and clinical assessment data at (2, 4 and ) 6 weeks post-treatment.

The study will evaluate whether serial serum measurements of galactomannan/beta-D-glucan during the first week(s) of antifungal therapy can distinguish between successful clinical outcome and failed clinical outcome at 6 weeks in patients with proven and probable invasive aspergillosis.

The study aims also at exploring various cut points for galactomannan/beta-D-glucan measurements at two weeks after initiation of antifungal therapy and at exploring the sensitivity and specificity for predicting clinical outcome at 6 and 12 weeks in patients with proven and probable invasive aspergillosis.

ELIGIBILITY:
Inclusion Criteria:

* proven or probable invasive aspergillosis with positive GM antigen test

Exclusion Criteria:

* Seronegative aspergillosis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hematology patients with proven or probable invasive aspergillosis
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-07; Primary Completion 2010-12 (Estimated); Study Completion 2011-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Johan A Maertens, MD, PhD, Principal Investigator — UZ Gasthuisberg Leuven